CLINICAL TRIAL: NCT01707628
Title: Response to Influenza Vaccination in Lymphoma Patients Treated With CHOP and Rituximab
Brief Title: Response to Influenza Vaccination in Lymphoma Patients Treated With Rituximab
Acronym: Rituxivac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, M. Rab, Drs., St. Antonius Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL37320.100.11
Record Dates: First submitted 2012-10-06; First posted 2012-10-16 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Non-Hodgkin Lymphoma (NHL)
Keywords: NHL; influenza vaccination; rituximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Influenza, Human | interventions — Influenza Vaccines; influvac; vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early group after rituximab (Active Comparator): Patients who received rituximab last dose 3-6 months before influenza vaccination will be the "early group".
  Interventions: Biological: influenza vaccination with influenza vaccine
- Late group after rituximab (Active Comparator): Patients who received rituximab last dose 9-12 months before influenza vaccination will be the "late group".
  Interventions: Biological: influenza vaccination with influenza vaccine
- Control group (Active Comparator): Healthy individuals will be receive vaccination with influenza vaccine and will serve as controls.
  Interventions: Biological: influenza vaccination with influenza vaccine

INTERVENTIONS:
Biological: influenza vaccination with influenza vaccine
  Other Names: Influvac; Vaxigrip

SUMMARY:
The purpose of this study is to compare the number of responders to vaccination with the influenza virus vaccine at different time points after last dose of rituximab in patients with lymphoma. Secondly to study the immune-response to vaccination with influenza virus vaccine, after treatment with rituximab in relation to the reconstitution of immune-function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-Hodgkin's lymphoma, treated with rituximab (with a range of 6-12 cycles) and who are in remission.
2. Completion of rituximab therapy in the last twelve months before start of the study.
3. Age ≥ 18 years.
4. Signing of informed consent.

Exclusion Criteria:

1. Completion of rituximab therapy 7-8 months before start of the study.
2. Fever at time of vaccination.
3. Previous/known allergic reaction to any of the components of the vaccines given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Influenza antibody titre | 3 weeks after vaccination

SECONDARY OUTCOMES:
number of memory B cells | 6 months
lymphocyte subsets | 6 months
immunoglobulin levels | 6 months
IgG subclasses | 6 months
production of IFN-γ by CD4+ cells | 6 months
Cytokines | 6 months
genetic factors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Minke AE Rab, Drs., Principal Investigator — St. Antonius Hospital
Locations (7):
- Netherlands (7):
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Onze Lieve Vrouwen Gasthuis, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overrijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Reinier de Graaf Groep, Delft, South Holland
  - Albert Schweitzer Hospital, Dordrecht, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht